CLINICAL TRIAL: NCT05531942
Title: Antiplatelet Effect of Ginkgo Diterpene Lactone Meglumine Injection in Acute Ischemic Stroke:A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Antiplatelet Effect of Ginkgo Diterpene Lactone Meglumine Injection in Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jm137312ccx
Record Dates: First submitted 2022-09-02; First posted 2022-09-08 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2022-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginkgo and aspirin (Active Comparator): Ginkgo Diterpene Lactone Meglumine Injection 25mg/5ml,once/day from Day 1 to Day 14. The injection was diluted with 250ml physiological saline,intravenous drip for about 3 hours;combined with Acetylsalicylic acid (Aspirin) given at a dose of 100 mg per day for 90 days.
  Interventions: Drug: Ginkgo Diterpene Lactone Meglumine Injection; Drug: Acetylsalicylic acid
- aspirin (Placebo Comparator): Patients in the aspirin group received the same volume saline injection as placebo for 14 days plus aspirin at a dose of 100 mg per day for 90 days.
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Ginkgo Diterpene Lactone Meglumine Injection — The injection was diluted with 250ml physiological saline,intravenous drip for about 3 hours.
  Other Names: YinxingErtieneizhiPu'an Zhusheye
  Arms: Ginkgo and aspirin
Drug: Acetylsalicylic acid — Acetylsalicylic acid (Aspirin) given at a dose of 100 mg/d for 90 days.
  Other Names: Aspirin

SUMMARY:
This study evaluates the addition of Ginkgo Diterpene Lactone Meglumine Injection to aspirin in the treatment of acute ischemic stroke.Half of patient will receive Ginkgo Diterpene Lactone Meglumine Injection(25mg once/day D1-D14) and aspirin(100mg once/day D1-D14) in combination, while the other half will receive aspirin(100mg once/day D1-D14).

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, placebo-controlled trial, A total of approximately 70 patients with acute ischemic stroke (5<NIHSS < 24), who can be treated within 4.5 to 48 hours of symptom onset will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive a Ginkgo Diterpene Lactone Meglumine Injection 25mg/5ml,once/day from Day 1 to Day 14(the injection was diluted with 250ml physiological saline,intravenous drip for about 3 hours), combined with Acetylsalicylic acid (Aspirin) at a dose of 100 mg/d for 90 days;2) the other group will receive the same volume saline injection as placebo for 14 days plus aspirin at a dose of 100 mg per day for 90 days.The primary objective is to assess the anti-platelet effects of Ginkgo Diterpene Lactone Meglumine Injection combined with Aspirin versus Aspirin alone in patients with acute ischemic stroke. The study consists of 3 visits including the day of randomization, Day 14±2days and Day 90±7days. The trial is anticipated to complete in 10 months from the first subject recruitment , with 70 subjects recruited. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Ethics Committee of Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS within 4.5-48 h of symptom onset;
* Age >40 years, and gender not limited;
* A score of 5-24 points on the National Institute of Health Stroke Scale (NIHSS);
* Written informed consent was available before enrolment.

Exclusion Criteria:

* Cardiogenic cerebral embolism;
* AIS caused by other definite causes (e.g., arterial dissection, vasculitis, vascular malformation, etc.) or undetermined etiology;
* Treated with thrombolysis or intravascular therapy, or with arteriovenous bridging after onset;
* Under dual antiplatelet therapy or anticoagulant therapy;
* A score of more than 2 on the modified Rankin Scale (mRS) (scores range from 0 [no symptoms] to 6 [death]) before the occurrence of AIS;
* Allergy or contraindication to GDLI or aspirin;
* Patients with active bleeding or bleeding tendency, malignancies, severe liver (the serum level of AST and/or ALT > 2 times the upper limit of normal), or renal failure (the serum level of creatinine > 1.5 times the upper limit of normal or GFR < 40 ml/min/1.73m2);
* Anticipated requirement for long-term nonstudy antiplatelet drugs or for nonsteroidal anti-inflammatory drugs affecting platelet function;
* Severe noncardiovascular coexisting condition, with a life expectancy of less than 3 months;
* Planned surgery or interventional treatment requiring cessation of the study drug;
* Pregnancy, lactation, or planning to get pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with NIHSS scores or NIHSS scores | 90 days
  Proportion of patients with National Institutes of Health Stroke Score (NIHSS) scores decrease ≥5 (Δ ≥ 5) or Modified Rankin Scale (mRS) scores decrease ≥2(Δ ≥ 2) from baseline to randomized 90 days.

SECONDARY OUTCOMES:
PL-11 AA at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of acetylsalicylic acid.
PL-11 ADP at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of adenosine diphosphate.
New vascular events defined as any event of the following: Any stroke (ischemic or hemorrhage) | 14 days
  All the new vascular events will be assessed by at least two neurologists based on neuroimaging and clinical feature. When there was disagreement, a third senior neurologist was consulted to reach a consensus decision.
PL-11 COL at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of collagen.
PL-11 EPI at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of epinephrine.

CONTACTS AND LOCATIONS:
Locations (1):
- Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No